CLINICAL TRIAL: NCT03449849
Title: Effect of Kale Consumption on Human Xenobiotic Metabolizing Enzymes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig Charron, Research Molecular Biologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS60 - Kale Study
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Base diet (Other): Subjects will consume a base diet prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Interventions: Other: Base Diet
- Kale Treatment (Other): Subjects will consume 500 g of kale per 2000 kcal of food, split between breakfast and dinner, as a supplement to the base diet.
  Interventions: Other: Kale Treatment

INTERVENTIONS:
Other: Base Diet — Base Diet
  Arms: Base diet
Other: Kale Treatment — Base Diet plus Kale
  Arms: Kale Treatment

SUMMARY:
The primary objective of this study is to determine how daily consumption of kale changes the activity of human xenobiotic metabolizing enzymes. Secondary objectives are to measure absorption and metabolism of kale phytonutrients, and to determine how kale consumption affects gene expression related to metabolism and lipid measures associated with cardiovascular health.

DETAILED DESCRIPTION:
Consumption of Brassica vegetables (which include broccoli, cabbage, and kale) is inversely associated with the incidence of several cancers, including cancers of the lung, stomach, liver, colon, rectum, breast, endometrium, and ovaries. Brassica vegetables are a good source of many nutrients, but the unique characteristic of Brassicas is their rich content of glucosinolates. Glucosinolates are sulfur-containing compounds that are converted to bioactive metabolites by a plant enzyme called myrosinase, which is released when the vesicles containing myrosinase are ruptured by chewing or cutting. These bioactive compounds are considered to be the active agent for cancer prevention. Their ability to reduce risk of cancer may derive in part from their ability to modulate foreign-substance metabolizing enzymes, which include enzymes called Phase I cytochrome P450s and Phase II enzymes.

The primary aim of this study is to investigate how daily consumption of kale influences foreign-substance metabolizing enzymes, which in turn may reduce cancer risk. Secondary aims of this study include measuring metabolism of kale nutrients, effect of kale consumption on fecal microbiota, and how kale consumption influences risk factors for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* 5 years cancer free
* Not a tobacco product user
* Blood glucose less than 126 mg/dL
* Able to voluntarily agree to participate and sign an informed consent document

Exclusion Criteria:

* Brassica vegetable allergy or intolerance
* use of oral contraceptives
* Women who have given birth in the previous 12 months
* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol, or Miradon (anisindione)
* History of bariatric surgery or nutrient malabsorption disease
* Pregnant, lactating, or intending to become pregnant during the study period
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
CYP1A2 activity will be analyzed | Day 7
  Plasma will be analyzed for caffeine metabolite ratios
CYP1A2 activity will be analyzed | Day 14
  Plasma will be analyzed for caffeine metabolite ratios
CYP1A2 activity will be analyzed | Day 42
  Plasma will be analyzed for caffeine metabolite ratios
CYP1A2 activity will be analyzed | Day 49
  Plasma will be analyzed for caffeine metabolite ratios.

SECONDARY OUTCOMES:
The ability of fecal microbiota to metabolize glucosinolates will be determined | Days 14 and 49.
  Fecal samples will be presented with glucosinolates to determine the change in the ability of fecal microbes to metabolize the glucosinolates.
Metabolites of Kale | On days 35 and 36
  Metabolites of Kale will be measured in plasma and urine.
Fecal microbiota will be analyzed for microbial DNA | Days 0, 14, 35, and 49
  Fecal microbial communities will be determined using DNA extracted from fecal samples.
UGT1A1 activity will be analyzed | On days 7, 14, 42, and 49
  Serum will be analyzed for bilirubin concentration to assess UGT1A1 activity
Glutathione S-transferase alpha concentration | On days 7, 14, 42, and 49
  Glutathione S-transferase alpha concentration will be measured in serum
Total cholesterol | On days 0, 7, 14, 35, 42, and 49
  Total cholesterol will be measured in serum
LDL cholesterol | On days 0, 7, 14, 35, 42, and 49
  LDL cholesterol will be measured in serum
HDL cholesterol | On days 0, 7, 14, 35, 42, and 49
  HDL cholesterol will be measured in serum
Triacylglycerides | On days 0, 7, 14, 35, 42, and 49
  Triacylglycerides will be measured in serum
Apolipoprotein A1 | On days 0, 7, 14, 35, 42, and 49
  Apolipoprotein A1 will be measured in serum
Apolipoprotein A2 | On days 0, 7, 14, 35, 42, and 49
  Apolipoprotein A2 will be measured in serum
Apolipoprotein B | On days 0, 7, 14, 35, 42, and 49
  Apolipoprotein B will be measured in serum
Changes in gene expression | On days 0, 14, 35, and 49
  messenger RNA concentrations in whole blood will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No